CLINICAL TRIAL: NCT06036550
Title: Inter- and Intra-observer Variability in First-trimester Uterine Artery Doppler Measurements.
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Wessel Ganzevoort, MD, PhD, Associate Professor, Gynaecologist-Perinatologist, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: uterine artery doppler
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Doppler Measurement of Uterine Artery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Doppler ultrasound measurement — Doppler sonographic assessment of the uterine artery was performed transabdominally. Patients underwent six sets of Doppler ultrasounds measurements of both right and left uterine artery.
  Other Names: Philips Ultrasound Inc. Bothell, WA, USA

SUMMARY:
The aim of this study is to investigate the inter- and intra-observer variability of first-trimester Uterine Artery Doppler ultrasound measurements in pregnancies between 11+0 and 13+0 weeks of gestation. Participants will undergo a measurement protocol (six sets of Doppler ultrasounds measurements of right and left uterine artery) performed alternately by two observers (sonographers or physicians who perform these ultrasounds frequently in clinical practice at the outpatient clinic).

DETAILED DESCRIPTION:
Doppler ultrasound measurements are increasingly performed in clinical practice to detect high-risk pregnancies. First-trimester uterine artery Doppler measurement might be a potential predictor for the development of maternal hypertensive disorders later on in pregnancy. However, before implementing this measurement into clinical practice and prediction models, the test characteristics of this first-trimester Doppler measurements should be adequately studied. The objective is to assess the inter- and intra-observer variability of first-trimester uterine Doppler ultrasound measurements.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Gestational age from 11+0 weeks to 13+6 weeks

Exclusion Criteria:

* Maternal age <18 years

  * Inability to give informed consent
  * Multiple pregnancy
  * Abnormal fetal heart tracings
  * Non-viable pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All women with a first-trimester singleton pregnancy receiving a Doppler ultrasound at the outpatient clinic are eligible.
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-04-06 (Actual)

PRIMARY OUTCOMES:
Inter- and intra-observer variability of first-trimester Uterine artery Doppler ultrasound | Between 11 and 13 weeks of gestation. Measurements will take place during general appointments and will take an extra 2-3 minutes
  The aim of this study is to investigate the inter- and intra-observer variability of first-trimester Uterine Artery Doppler ultrasound measurements, according to the TRUST-study criteria for reproducibility assessment and analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam University Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Coelho Neto MA, Roncato P, Nastri CO, Martins WP. True Reproducibility of UltraSound Techniques (TRUST): systematic review of reliability studies in obstetrics and gynecology. Ultrasound Obstet Gynecol. 2015 Jul;46(1):14-20. doi: 10.1002/uog.14654. Epub 2015 Jun 4. PMID 25175693
- [Background] Khalil A, Nicolaides KH. How to record uterine artery Doppler in the first trimester. Ultrasound Obstet Gynecol. 2013 Oct;42(4):478-9. doi: 10.1002/uog.12366. Epub 2013 May 8. No abstract available. PMID 23658028
- [Result] Marchi L, Zwertbroek E, Snelder J, Kloosterman M, Bilardo CM. Intra- and inter-observer reproducibility and generalizability of first trimester uterine artery pulsatility index by transabdominal and transvaginal ultrasound. Prenat Diagn. 2016 Dec;36(13):1261-1269. doi: 10.1002/pd.4970. Epub 2016 Dec 6. PMID 27862084